CLINICAL TRIAL: NCT04419896
Title: The Informed Genetics Annotated Patient Registry: The iGAP Registry
Brief Title: The Informed Genetics Annotated Patient Registry
Acronym: iGAP
Status: Enrolling by invitation | Type: Observational
Sponsor: Medneon (Industry)
Responsible Party: Sponsor
Other Study IDs: IGAP1000
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Predisposition, Genetic
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Inclusion criteria for Retrospective Subjects:
  * Men and women 18 years or older;
  * Is or was a patient of a Participating Practice and was previously tested with Germline, Genomic, or other Biomarker Tests; and
  * For Germline Genetic Test patients, have a diagnosis of cancer or pathogenic or likely pathogenic (P/LP) result.
- Prospective: Inclusion criteria for Prospective Subjects:
  * Men and women aged 18 years or older;
  * Presents consecutively to a Participating Practice and who has previously been screened and tested (i.e., is a new patient scheduled for a visit at a Participating Practice or is an existing patient who returns to a Participating Practice);
  * Receives or has received Germline, Genomic, or other Biomarker Testing, either through a prior healthcare provider or a Participating Practice; and
  * Consents to be a part of the Registry.

SUMMARY:
This prospective and retrospective registry will evaluate the clinical effectiveness of Germline Genetic, Genomic, and other Biomarker testing results over time in different clinical populations, in order to shape guidelines for testing, patient management, and precision therapy.

DETAILED DESCRIPTION:
Interest and knowledge about the genetics and biology of an individual's inherited risk of disease and progression of disease is growing. Physicians are increasing using tests and technology, including Germline Genetic, Genomic, and Biomarker Testing, to provide insight into a healthy individual's risk and an affected individual's disease characteristics, in order to provide individualized clinical treatments. However, many barriers to widespread and appropriate Germline Genetic, Genomic, and Biomarker Testing persist due to complex guidelines for use, varied quality and cost, rapid advances, and adequate understanding of appropriate implementation by medical professionals. The iGAP Registry is a multi-center ongoing database designed to capture information on disease risk assessment, Germline Genetic, Genomic, and Biomarker Testing, and their utilization and impact on treatment practices and outcomes to help determine, over time, the most effective use of testing in varied patient populations and to support the increased use of precision medicine.

ELIGIBILITY:
Inclusion Criteria for Retrospective Subjects:

* Men and women 18 years or older;
* Is or was a patient of a Participating Practice and was previously tested with Germline, Genomic, or other Biomarker Tests; and
* For Germline Genetic Test patients, have a diagnosis of cancer or pathogenic or likely pathogenic (P/LP) result.

Inclusion Criteria for Prospective Subjects:

* Men and women aged 18 years or older;
* Presents consecutively to a Participating Practice and who has previously been screened and tested (i.e., is a new patient scheduled for a visit at a Participating Practice or is an existing patient who returns to a Participating Practice);
* Receives or has received Germline, Genomic, or other Biomarker Testing, either through a prior healthcare provider or a Participating Practice; and
* Consents to be a part of the Registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years or older who meet eligibility criteria, who is screened and tested for or receives or has received Germline, Genomic, or other Biomarker Testing.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
To understand the utilization of Germline Genetic, Genomic, and Biomarker Testing in various clinical settings. | 10 years
  To understand the utilization of Germline Genetic, Genomic, and Biomarker Testing in various clinical settings. The registry will gather information on patient demographics and personal and family history, as well as test results of Germline Genetic, Genomic, and Biomarker tests.

SECONDARY OUTCOMES:
To understand Physician Decision Impact and Patient Reported Outcomes resulting from the utilization of Germline Genetic, Genomic, and Biomarker testing. | 10 years
  To understand Physician Decision Impact and Patient Reported Outcomes resulting from the utilization of Germline Genetic, Genomic, and Biomarker testing. This registry will gather information to capture the clinical management decision making processes of the physicians, before and after receiving information from Germline Genetic, Genomic, or other Biomarker testing. Further, this registry will collect information on Patient Reported Outcomes, or patient described impacts of Germline Genetic, Genomic, or other Biomarker testing on their treatment, clinician interactions, follow-up, and mental health.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - North Valley Breast Clinic, Redding, California
  - Advocate Good Shepherd, Barrington, Illinois
  - Comprehensive Breast Care, Troy, Michigan
  - Nashville Breast Center, Nashville, Tennessee
  - Dallas Surgical, Dallas, Texas